CLINICAL TRIAL: NCT03664895
Title: Density Lowering Effect of Ovarian Function Suppression in Premenopausal Breast Cancer Patients Who Had no Density Change With One Year of Tamoxifen Treatment
Brief Title: Density Lowering Effect of "OFS Add on to TMX"(DELFINO Trial)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DELFINO trial
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer Invasive
Keywords: premenopausal women, MMG density, Ovary function suppression
MeSH Terms: interventions — Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- observation arm(TMX, MDR≥5%) (No Intervention): keep go on TMX
- control arm(TMX, MDR<5%) (No Intervention): keep go on TMX
- OFS add arm(TMX + OFS, MDR<5%) (Active Comparator): OFS add on to TMX
  Interventions: Drug: Leuplin or zoladex

INTERVENTIONS:
Drug: Leuplin or zoladex — OFS(Leuplin or zoladex) add on to TMX
  Arms: OFS add arm(TMX + OFS, MDR<5%)

SUMMARY:
DELFINO tial is designed to investigate the role of "OFS add on to TMX ", based on MMG density as a surrogate marker in premenopausal women

* Premise - MMG density as a surrogate marker of hormone therapy
* Assumption - "Add on OFS to TMX" would have further decrease of density

  * 3-arm(Observation arm + Randomised 2-arm), phase III, RCT with 1:1 allocation

DETAILED DESCRIPTION:
Enroll : Sep03,2018~(Planned N= 224)

1. Inclusion criteria

   * Premenopausal
   * ER+
   * Planned tamoxifen(TMX)
   * No planned ovary function suppression(OFS)
   * Regardless of ChemoTx
   * Mammography(MMG) density check via Volpara*(=Baseline MMG density, BaMD) (*Volpara= software to check MMG density)
2. Check MMG Density via Volpara After 1yr TMX (At1yrMD) Check menopausal status after 1yr TMX(Menstruation episode or FSH <30)
3. MMG Density Reduction(MDR =BaMD-AtMD ) at 1yr
4. MDR ≥5% -> Keep go on TMX MDR <5% -> 1:1 randomization -> Keep go on TMX vs OFS add on to TMX
5. Analysis : 5yr MDR (1'endpoint), 5yr DFS(2'endpoint), 5yr OS
6. Calculation of patients' number In previous study(<Kim et al. Breast Can Res 2012>) MDR (Mammography Density Reduction) was found in about 50% of all patients who received endocrine therapy.

Expected

* MDR in "TMX only" cohort -> 6 ± 7%
* MDR in "OFS add on to TMX" -> 10 ± 7%

  * after 1yr, Significance level 5%, average MDR 4% difference, 80% power, 10% dropout rate => 1:1 randomization Number = 112(56:56) Total number = 224

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women, ER+ breast cancer, stage I~III, underwent standard treatment including surgery, Planned TMX
* available MMG density check via Volpara

Exclusion Criteria:

* Bilateral breast cancer
* Prior endocrine therapy
* Postmenopausal status
* unavailable MMG density check via volpara before and after TMX

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 224 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MMG density Reduction | 5 years

SECONDARY OUTCOMES:
Disease free survival | 5 years

OTHER OUTCOMES:
overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Wonshik Han, Study Chair — Seoul National University College of Medicine/Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided